CLINICAL TRIAL: NCT07307677
Title: Effect of Melatonin and Metformin Combination Therapy on Clinical and Biochemical Parameters inInsulin Resistant Polycystic Ovary Syndrome Compared to Metformin Alone
Brief Title: Melatonin & Metformin on Clinical & Biochemical Parameters in Insulin Resistant PCOS Compared to Metformin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mst.Sumyara Khatun (Other)
Collaborators: Bangladesh Medical University (Other)
Responsible Party: Sponsor-Investigator, Mst.Sumyara Khatun, Medical Officer, Bangladesh Medical University
Organization: Bangladesh Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5498
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: PCOS(Insulin Resistant)
Keywords: Melatonin in PCOS
MeSH Terms: interventions — Metformin; Melatonin

STUDY DESIGN:
Intervention Model Description: Open label parallel design randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: Melatonin and Metformin (Experimental): Participants will receive Melatonin (3mg) 3 tablet single dose at night for 12 weeks and Metformin (500mg) once daily for 7days followed by twice daily for next 7 days followed by thrice daily for next 10 weeks
  Interventions: Combination Product: Melatonin 3mg
- Comparator arm: Metformin (Active Comparator): Participants will receive Metformin (500mg) once daily for 7days followed by twice daily for next 7 days followed by thrice daily for next 10 weeks
  Interventions: Drug: Metformin 500mg

INTERVENTIONS:
Drug: Metformin 500mg — Metformin (500mg) once daily for 7days followed by twice daily for next 7 days followed by thrice daily for next 10 weeks
  Arms: Comparator arm: Metformin
Combination Product: Melatonin 3mg — Melatonin (3mg) 3 tablet single dose at night for 12 weeks and Metformin (500mg) once daily for 7days followed by twice daily for next 7 days followed by thrice daily for next 10 weeks
  Arms: Experimental arm: Melatonin and Metformin

SUMMARY:
Women with polycystic ovary syndrome with HOMA-IR >2.6 fulfilling inclusion and exclusion criteria will be randomly allocated into two groups:experimental group: A (Melatonin 3mg and Metformin 500mg) and control group: B (Metformin 500mg). Each group will be contained 30 selected patients.

Group B:Tab. Metformin (500mg) once daily for 7days followed by twice daily for next 7 days followed by thrice daily for next 10 weeks.

Outcome variables will be measured after three months, will be meticulously recorded for analysis and comparison.

DETAILED DESCRIPTION:
After obtaining approval of the Institutional Review Board (IRB), this randomized controlled trial will be conducted at Bangabandhu Sheikh Mujib Medical University (BSMMU). Already diagnosed patients of polycystic ovary syndrome with subfertility with HOMA-IR >2.6 attending in the OPD of Reproductive Endocrinology and Infertility department at BSMMU will be the study population. Women with PCOS fulfilling inclusion and exclusion criteria will be explained in details regarding the objectives, rationality, procedure and potential benefits of the study. The patients will be counselled regarding the drugs and side effects and Informed written consent will be obtained before enrollment.Random allocation will be done using serially numbered closed opaque envelopes. Eligible women will be randomly allocated into two groups:experimental group: A and control group: B. Each group will be contained 30 selected patients.

Group A:Tab. Melatonin (3mg) 3 tablet once daily at night for 12 weeks with Tab. Metformin (500mg) once daily for 7days followed by twice daily for next 7 days followed by thrice daily for next 10 weeks.

Group B:Tab. Metformin (500mg) once daily for 7days followed by twice daily for next 7 days followed by thrice daily for next 10 weeks.

Data will be collected through interviews, physical examinations and laboratory investigations. Prior to commencement of treatment, full assessments including demographic and clinical information and the result of baseline investigations will be undertaken.

Follow up: Participants will come after one month to assess compliance with the regimen and monitor for any potential side effects. A third visit will be scheduled at the end of the third month for a comprehensive assessment. Any adverse events experienced by participants will be carefully noted and documented throughout the study duration. Outcome variables will be measured after three months, will be meticulously recorded for analysis and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed case of PCOS according to Rotterdam criteria
* Women of age 18-35 years
* Insulin resistance (HOMA-IR >2.6)

Exclusion Criteria:

* BMI: ≤ 18.5 and ≥ 30 kg/m2
* Uncontrolled endocrine disorders (Diabetis melitus, Hypothyroidism, Hyperprolactinemia)
* Known case of any medical disease (Renal, hepatic or cardiac disease)
* Any medication which would affect insulin resistance (Metformin, Myo- inositol, Pioglitazone) in last three months.
* Hypersensitivity to melatonin.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline to 12 weeks
  HOMA-IR calculated by the following formula:
  HOMA-IR= Fasting glucose (mmol/L) x Fasting insulin mIU/ml divided by 22.5. For the present study HOMA-IR >2.6 can be considered as insulin resistance

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline to 12 weeks
  Body mass index is calculated by dividing the weight in kg by the height in meter square to assess obesity
Change in Waist Circumference | Baseline to 12 weeks
  Waist Circumference is measured in centimeter by placing a tape horizontally midway between the lower border of ribs and iliac crest on the mid axillary line.

CONTACTS AND LOCATIONS:
Overall Officials: Jesmine Banu, MS, Study Chair — Bangladesh Medical University; Farzana Rahman, MBBS, Principal Investigator — Bangladesh Medical University
Locations (1):
- Bangladesh Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Zhang H, Guo B, Tao Y, Zhang J, Wang J, Chen G, Cheng M, Hong Q, Cao Y, Xie F. Melatonin refines ovarian mitochondrial dysfunction in PCOS by regulating the circadian rhythm gene Clock. Cell Mol Life Sci. 2025 Mar 6;82(1):104. doi: 10.1007/s00018-025-05609-9. PMID 40047877
- [Background] Ziaei S, Hasani M, Malekahmadi M, Daneshzad E, Kadkhodazadeh K, Heshmati J. Effect of melatonin supplementation on cardiometabolic risk factors, oxidative stress and hormonal profile in PCOS patients: a systematic review and meta-analysis of randomized clinical trials. J Ovarian Res. 2024 Jul 4;17(1):138. doi: 10.1186/s13048-024-01450-z. PMID 38965577